CLINICAL TRIAL: NCT03410056
Title: A Phase 1b/2a Study to Evaluate the Safety and Efficacy of Efavaleukin Alfa in Subjects With Active Rheumatoid Arthritis With Inadequate Response to Standard of Care Therapy
Brief Title: Safety and Efficacy of Efavaleukin Alfa in Subjects With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Amgen made a business decision not to proceed with Phase 2.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20170149; 2017-001944-36 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-25 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis RA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1b: Placebo (Placebo Comparator): Matching placebo administered via subcutaneous injection for a total of up to 12 weeks. Participants received placebo in 1 of 2 dosing schedules (i.e. dosing schedule A [less frequent] or schedule B [more frequent]).
  Interventions: Drug: Placebo
- Phase 1b: Efavaleukin alfa Cohort 1 (Experimental): A low dose of Efavaleukin alfa administered via subcutaneous injection using dosing schedule A (less frequent than schedule B) for a total of up to 12 weeks.
  Interventions: Drug: Efavaleukin alfa
- Phase 1b: Efavaleukin alfa Cohort 2 (Experimental): A high dose of Efavaleukin alfa administered via subcutaneous injection using dosing schedule A (less frequent than schedule B) for a total of up to 12 weeks.
  Interventions: Drug: Efavaleukin alfa
- Phase 1b: Efavaleukin alfa Cohort 3 (Experimental): A medium dose of Efavaleukin alfa administered via subcutaneous injection using dosing schedule B (more frequent than schedule A) for a total of up to 12 weeks.
  Interventions: Drug: Efavaleukin alfa
- Phase 1b: Efavaleukin alfa Cohort 4 (Experimental): A medium/high dose of Efavaleukin alfa administered via subcutaneous injection using dosing schedule B (more frequent than schedule A) for a total of up to 12 weeks.
  Interventions: Drug: Efavaleukin alfa
- Phase 2a: Placebo (Placebo Comparator): Matching placebo administered via subcutaneous injection, depending on the recommended phase 2 dose (RP2D) and dosing schedule as determined in phase 1b, for a total of up to 12 weeks.
  Interventions: Drug: Placebo
- Phase 2a: Efavaleukin alfa (Experimental): Efavaleukin alfa administered via subcutaneous injection depending on the RP2D and dosing schedule determined in phase 1b, for up to a total of up to 12 weeks.
  Interventions: Drug: Efavaleukin alfa

INTERVENTIONS:
Drug: Efavaleukin alfa — Efavaleukin alfa administered as a subcutaneous injection.
  Other Names: AMG 592
  Arms: Phase 1b: Efavaleukin alfa Cohort 1; Phase 1b: Efavaleukin alfa Cohort 2; Phase 1b: Efavaleukin alfa Cohort 3; Phase 1b: Efavaleukin alfa Cohort 4; Phase 2a: Efavaleukin alfa
Drug: Placebo — Placebo administered as a subcutaneous injection.
  Arms: Phase 1b: Placebo; Phase 2a: Placebo

SUMMARY:
Phase 1b. To evaluate the safety and tolerability of subcutaneous (SC) dose administrations of Efavaleukin alfa in subjects with active rheumatoid arthritis (RA).

Phase 2a. To evaluate the efficacy of Efavaleukin alfa at week 12 as measured by the American College of Rheumatology 20 percent improvement criteria (ACR 20) in adult subjects with moderate to severe RA.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 to ≤ 70 years of age at screening.
* A diagnosis of RA consistent with the 1987 or 2010 American College of Rheumatology (ACR)/European League Against Rheumatism classification criteria.
* Active RA defined as: Phase 1b: DAS-28-CRP > 2.6 at screening. The 28-joint count consists of the finger joints excluding the distal interphalangeal joints, the wrists, elbows, shoulders, and knees. Phase 2a: ≥ 6 swollen joints (based on 66-joint count) and ≥ 6 tender joints (based on 68-joint count) at screening and baseline. The distal interphalangeal joint should be evaluated but not included in the total count to determine eligibility. Additionally, C-reactive protein (CRP) must be greater than the upper limit of normal (ULN) per the central laboratory at screening.
* Receiving treatment with methotrexate for ≥ 12 weeks and on a stable dose ≥ 15 mg weekly for ≥ 8 weeks prior to day 1. A lower methotrexate dose is acceptable (but no lower than 10 mg weekly) if it is the highest tolerated dose and gastrointestinal or hematologic toxicity at doses ≥ 15 mg weekly is documented by the investigator.
* Receiving treatment with folic or folinic acid per investigator judgment or according to local standard of care.
* Phase 1b only: Subject may be receiving a stable dose of leflunomide, sulfasalazine, hydroxychloroquine, minocycline in combination with methotrexate and the dose must be stable for ≥ 8 weeks prior to day 1.
* Subject may be receiving a stable dose of prednisone ≤ 10mg daily or other equivalent corticosteroid dose and the dose must be stable for ≥ 2 weeks prior today 1.
* Phase 1b only. Normal or clinically acceptable electrocardiogram (ECG) values (12-lead reporting ventricular rate and PR, QRS, QT and QTc interval) at screening and baseline based on opinion of the investigator.
* Immunizations (tetanus, diphtheria, pertussis, seasonal influenza [during flu season], and pneumococcal [polysaccharide] vaccinations) up to date per local standards as determined by the investigator.

Exclusion Criteria:

* Class IV RA according to ACR revised response criteria
* Diagnosis of Felty's Syndrome (RA, splenomegaly and granulocytopenia).
* Prosthetic joint infection within 3 years of screening or native joint infection within 1 year prior to screening.
* Active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to day 1 OR presence of serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to day 1.
* Known history of active tuberculosis.
* Positive test for tuberculosis during screening defined as either: positive purified protein derivative (PPD) (≥ 5 mm of induration at 48 to 72 hours after test is placed) OR positive Quantiferon test: a positive PPD and a history of Bacillus Calmette-Guérin vaccination are allowed with a negative Quantiferon test and negative chest x ray; a positive PPD test (without a history of Bacillus Calmette-Guérin vaccination) or a positive or indeterminate Quantiferon test are allowed if they have ALL of the following at screening: no symptoms per tuberculosis or sheet provided by Amgen; document history of a completed course of adequate prophylaxis(completed treatment for latent tuberculosis per local standard of care prior to the start of investigational product); no known exposure to a case of active tuberculosis after most recent prophylaxis; negative chest X-ray.
* Positive for hepatitis B surface antigen, hepatitis B core antibody (confirmed by hepatitis B deoxyribonucleic acid (DNA) polymerase chain reaction [PCR] test) or detectable hepatitis C virus ribonucleic acid (RNA) by PCR (screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive). A history of hepatitis B vaccination without history of hepatitis B is allowed.
* Phase 1b only: Positive for Human Immunodeficiency Virus (HIV) at screening or known to be HIV positive. Phase 2a only: Known history of HIV
* Phase 1b only: Positive drug or alcohol urine test for illicit drugs at screening. Prescription medications detected by the drug test are allowed if they are being taken under the direction of a physician.
* Presence of one or more significant concurrent medical conditions per investigator judgment, including but not limited to the following: poorly controlled diabetes or hypertension; chronic kidney disease stage IIIb, IV, or V; symptomatic heart failure (New York Heart Association class II, III, or IV); myocardial infarction or unstable angina pectoris within the past 12 months prior to randomization; severe chronic pulmonary disease (eg, requiring oxygen therapy); multiple sclerosis or any other demyelinating disease; major chronic inflammatory disease or connective tissue disease other than RA (eg, systemic lupus erythematosus with the exception of secondary Sjögren's syndrome).
* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years.
* History of alcohol or substance abuse within 6 months of screening
* Phase 1b only: Current smoker, and/or use of any nicotine or tobacco containing products within the last 6 months prior to day 1. These types of products include but are not limited to: snuff, chewing tobacco, cigars, electronic cigarettes, cigarettes, pipes, or nicotine patches.
* Phase 1b only: Subject unwilling to limit alcohol consumption to ≤ 1 drink of alcohol per day and ≤ 3 drinks per week for the duration of the study, where a drink is equivalent to 12 ounces of regular beer, 8 to 9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits. Phase 1b only: Unwilling or unable to abstain from alcohol consumption within 48 hours prior to each visit (including screening).
* Subjects who have received intra-articular or systemic corticosteroid injections for treatment of acute RA flare (not being part of a regular therapeutic regimen) within 4 weeks prior to screening.
* Currently receiving or had treatment with cyclophosphamide, chlorambucil, nitrogen mustard, or any other alkylating agent ≤ 6 months prior to day 1.
* Prior treatment with more than a total of 3 therapies that include biologic disease modifying anti-rheumatic drug (DMARDs) or oral synthetic DMARDs (such as tofacinitib, baricitinib). Prior treatment consists of at least 4 doses of a given therapy where the doses were given solely for treatment of RA disease. Prior therapies must not have been used within the following time periods:

  * ≤ 4 weeks prior to day 1 for etanercept and anakinra
  * ≤ 6 months for rituximab
  * ≤ 2 weeks for oral janus kinase inhibitors
  * ≤ 9 weeks prior to day 1 for all therapies not listed above
* Currently receiving or had treatment with any of the following ≤ 12 weeks prior to day 1:

  * azathioprine
  * cyclosporine
  * gold
  * mycophenolate mofetil
  * Prosorba column
  * Tacrolimus
* Phase 2a only: Currently receiving or had treatment with leflunomide ≤ 12 weeks prior to day 1 unless an active washout with cholestyramine has been performed.
* Phase 2a only: Currently receiving or had treatment with any of the following ≤ 4 weeks prior to day 1:

  * hydroxychloroquine
  * sulfasalazine
  * minocycline
  * oral janus kinase inhibitor (eg, tofacitinib, baricitinib)
  * intra-articular, intramuscular or intravenous corticosteroids, including adrenocorticotropic hormone
  * intra-articular hyaluronic acid injections
  * live vaccines -- For Phase 2 only:
* Unstable dose of non-steroidal anti-inflammatory drugs (NSAID), acetaminophen, and/or analgesics which is taken on an unscheduled basis (ie, not daily or scheduled every certain number of hours) and/or initiated <4 weeks prior to day 1.
* Received the following within 12 hours prior to screening or day 1:

acetaminophen, NSAIDs, tramadol, and/or any narcotic analgesics such as but not limited to hydrocodone, codeine, tramadol, propoxyphene and/or oxycodone (unless in the form of oxycontin). Subject has taken oxycontin within 24 hours prior to screening or day 1.

* Phase 1b only: Received any herbal medicines (eg St John's wort),or non-vitamin dietary supplements (eg, magnesium) with the exception of calcium within 4 weeks prior to day 1.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Presence of laboratory abnormalities at screening including the following:

  * Aspartate aminotransferase (AST) or alanine amino transferase (ALT) at screening > 1.5X upper limit of normal (ULN)
  * Serum total bilirubin (TBL) ≥ 1.5 mg/dL (≥ 26 μmol/L)
  * Hemoglobin ≤ 10.5 g/dL(≤105 g/L)
  * Platelet count < 100,000/mm^3 (<100 x 10^9/L)
  * White blood cell count < 2,500 cells/mm^3 (2.5 x 10^9/L)
  * Absolute neutrophil count (ANC) < 1,000/mm^3 (1.0 x 10^9/L)
  * Calculated glomerular filtration rate of ≤ 50 mL/min/1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula
* Any other laboratory abnormality, which, in the opinion of the investigator, poses a safety risk, will prevent the subject from completing the study, will interfere with the interpretation of the study results, or might cause the study to be detrimental to the subject.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 weeks after the last dose of investigational product.
* Females of child-bearing potential with a positive pregnancy test (assessed by a serum pregnancy test at screening and a urine pregnancy test at baseline).
* Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 6 weeks after the last dose of investigational product.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments [COAs]) to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (5):
  - Research Site, Anniston, Alabama
  - Research Site, Torrance, California
  - Research Site, Lansing, Michigan
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas
- Research Site, Sofia, Bulgaria
- Germany (2):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
- Poland (6):
  - Research Site, Józefów
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Stalowa Wola
  - Research Site, Świdnik
  - Research Site, Wroclaw
- Research Site, A Coruña, Galicia, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in phase 1b were to be enrolled into 1 of 4 planned dosing cohorts and randomized in a 3:1 ratio to receive Efavaleukin alfa or placebo according to 1 of 2 dosing schedules; A (less frequent) and B (more frequent).
Pre-assignment Details: Enrollment of the phase 1b part of this study was stopped as of 30 September 2019, due to data that suggested that there is not sufficient benefit-risk for the use of Efavaleukin alfa plus standard of care therapy in this study population. The study was terminated prior to the enrollment of any participants into phase 1b Cohort 4 and phase 2a cohorts.
Groups:
- Phase 1b: Efavaleukin Alfa Cohort 4: A medium/high dose of Efavaleukin alfa administered via subcutaneous injection using dosing schedule B (more frequent than schedule A) for a total of up to 12 weeks.
  No participants were enrolled into this cohort as the study was terminated prior to initiation of Cohort 4.
- Phase 2a: Placebo: Matching placebo administered via subcutaneous injection, depending on the recommended phase 2 dose (RP2D) and dosing schedule as determined in phase 1b, for a total of up to 12 weeks.
  The study was terminated prior to the start of phase 2a and no participants were enrolled.
- Phase 2a: Efavaleukin Alfa: Efavaleukin alfa administered via subcutaneous injection depending on the RP2D and dosing schedule determined in phase 1b, for up to a total of up to 12 weeks.
  The study was terminated prior to the start of phase 2a and no participants were enrolled.
Period: Overall Study
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3 | Phase 1b: Efavaleukin Alfa Cohort 4 | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Started | 8 | 6 | 11 | 11 | 0 | 0 | 0
Received Treatment | 8 | 6 | 11 | 11 | 0 | 0 | 0
Completed | 8 | 4 | 3 | 6 | 0 | 0 | 0
Not Completed | 0 | 2 | 8 | 5 | 0 | 0 | 0
Not completed — Decision by Sponsor | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 5 | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set: All participants who received at least 1 dose of investigational product.
  Only cohorts with enrolled participants are included in the baseline population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3 | Total
Number analyzed (Participants) | 8 | 6 | 11 | 11 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.1) | 57.8 (8.4) | 53.1 (10.7) | 51.4 (15.3) | 51.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 9 | 8 | 27
  Male | 4 | 0 | 2 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 4
  Not Hispanic or Latino | 7 | 6 | 9 | 10 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 6 | 5 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were events with an onset after the administration of the first dose of study treatment.
  TEAEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE).
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limited age appropriate instrumental activities of daily life (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling; limited self care ADL.
  Grade 4 Life-threatening consequences; urgent interventions indicated.
  Serious adverse events (SAEs) were defined as meeting at least 1 of the following criteria:
  * Results in death (fatal)
  * Immediately life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other medically important serious event
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: The safety analysis set: All participants who received at least 1 dose of investigational product. Only cohorts with enrolled participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 6 | 11 | 11
Participants
  TEAEs | 3 | 5 | 11 | 11
  Grade ≥ 2 TEAEs | 2 | 3 | 8 | 8
  Grade ≥ 3 TEAEs | 0 | 0 | 1 | 0
  Grade ≥ 4 TEAEs | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 1 | 0
  TEAEs leading to discontinuation of study treatment | 0 | 1 | 7 | 3
  Life-threatening TEAEs | 0 | 0 | 0 | 0
  Fatal TEAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Clinically Significant Change in Vital Signs
Description: Any changes in systolic/diastolic blood pressure, heart rate, respiratory rate, and temperature that were deemed as clinically significant by the Investigator were reported.
Time Frame: Baseline up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 6 | 11 | 11
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Clinically Significant Change in Laboratory Safety Tests
Description: Laboratory safety tests included chemistry and hematology parameters. Clinically significant laboratory safety tests were any events assessed as CTCAE Grade ≥3 at any post-baseline visit.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling; limited self care ADL.
  Grade 4 Life-threatening consequences; urgent interventions indicated.
Time Frame: Baseline up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 6 | 11 | 11
Participants | 0 | 0 | 1 | 0

4. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Clinically Significant Change in Electrocardiograms (ECGs)
Description: Any changes in ECG parameters that were deemed clinically significant by the investigator were reported.
Time Frame: Baseline up to end of treatment maximum of 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 6 | 11 | 11
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Phase 2a: Number of Participants Who Achieved an American College of Rheumatology 20 Percent Improvement Criteria (ACR 20) at Week 12
Description: ACR 20 response defined as at least 20 percent improvement from baseline in both tender and swollen joint counts, and a 20 percent improvement or more in at least 3 of the following 5 criteria:
  * physician global assessment of disease activity (PGA)
  * subject global assessment of disease activity (SGA)
  * patient global assessment of joint pain
  * subject self-assessment of disability (HAQ-DI)
  * C-Reactive Protein (CRP)
Time Frame: Baseline and Week 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 1b: Efavaleukin Alfa Serum Concentrations
Description: A summary of mean serum concentrations of Efavaleukin alfa over time is presented. Any results below the lower limit of quantification were set to 0.00.
Time Frame: Day 1 (pre-dose), 6 and 12 hours post-dose, and days 2, 3, 4, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, and Day 85 (pre-dose), 6 and 12 hours post-dose and days 86, 87, 88, 92, 99, 113 and 127
Population: The pharmacokinetic (PK) analysis set: All participants who received at least one dose of Efavaleukin alfa and had at least one quantifiable PK sample collected. Only participants with PK data available for analysis are presented. Only cohorts with enrolled participants are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 6 | 11 | 11
ng/mL
  Day 1 (pre-dose) | 0.00 (0.00) | 0.0 (0.00) | 0.00 (0.00)
  Day 1 (6 hours post-dose) | 1.35 (0.795) | 7.67 (8.01) | 2.13 (2.98)
  Day 1 (12 hours post-dose) | 2.43 (0.867) | 14.6 (12.1) | 4.09 (4.70)
  Day 2 | 2.59 (0.875) | 22.0 (11.5) | 5.44 (5.09)
  Day 3 | 1.70 (0.850) | 18.6 (9.16) | 3.65 (3.13)
  Day 4: number analyzed (Participants) | 6 | 11 | 9
  Day 4 | 0.727 (0.277) | 7.65 (5.85) | 2.36 (2.84)
  Day 8: number analyzed (Participants) | 6 | 10 | 10
  Day 8 | 0.0555 (0.0924) | 0.108 (0.146) | 0.0284 (0.0624)
  Day 11: number analyzed (Participants) | 5 | 10 | 10
  Day 11 | 0.0230 (0.0514) | 0.0115 (0.0364) | 0.930 (0.780)
  Day 15: number analyzed (Participants) | 5 | 8 | 8
  Day 15 | 0.00 (0.00) | 0.00 (0.00) | 0.107 (0.150)
  Day 22: number analyzed (Participants) | 3 | 6 | 7
  Day 22 | 0.0830 (0.144) | 0.0703 (0.112) | 0.235 (0.373)
  Day 29: number analyzed (Participants) | 3 | 6 | 7
  Day 29 | 0.00 (0.00) | 0.00 (0.00) | 0.217 (0.344)
  Day 36: number analyzed (Participants) | 5 | 4 | 8
  Day 36 | 0.0644 (0.144) | 0.102 (0.203) | 0.239 (0.425)
  Day 43: number analyzed (Participants) | 5 | 4 | 7
  Day 43 | 0.00 (0.00) | 0.00 (0.00) | 0.104 (0.275)
  Day 50: number analyzed (Participants) | 4 | 4 | 7
  Day 50 | 0.205 (0.304) | 0.105 (0.210) | 0.122 (0.322)
  Day 57: number analyzed (Participants) | 4 | 4 | 7
  Day 57 | 0.0368 (0.0735) | 0.00 (0.00) | 0.0886 (0.234)
  Day 64: number analyzed (Participants) | 2 | 4 | 5
  Day 64 | 0.336 (NA) — Insufficient samples were collected to assess SD. | 0.212 (0.424) | 0.0294 (0.0657)
  Day 71: number analyzed (Participants) | 2 | 4 | 5
  Day 71 | 0.0635 (NA) — Insufficient samples were collected to assess SD. | 0.00 (0.00) | 0.00 (0.00)
  Day 78: number analyzed (Participants) | 3 | 4 | 6
  Day 78 | 0.154 (0.267) | 0.355 (0.614) | 0.0508 (0.0819)
  Day 85 (pre-dose): number analyzed (Participants) | 4 | 3 | 6
  Day 85 (pre-dose) | 0.00 (0.00) | 0.00 (0.00) | 0.0578 (0.0958)
  Day 85 (6 hours post-dose): number analyzed (Participants) | 4 | 2 | 6
  Day 85 (6 hours post-dose) | 2.41 (1.56) | 5.91 (NA) — Insufficient samples were collected to assess SD. | 1.92 (2.64)
  Day 85 (12 hours post-dose): number analyzed (Participants) | 4 | 2 | 6
  Day 85 (12 hours post-dose) | 4.00 (2.05) | 12.9 (NA) — Insufficient samples were collected to assess SD. | 2.92 (4.03)
  Day 86: number analyzed (Participants) | 4 | 2 | 6
  Day 86 | 3.60 (2.07) | 12.3 (NA) — Insufficient samples were collected to assess SD. | 2.97 (4.48)
  Day 87: number analyzed (Participants) | 4 | 2 | 6
  Day 87 | 2.10 (1.15) | 4.39 (NA) — Insufficient samples were collected to assess SD. | 1.87 (2.43)
  Day 88: number analyzed (Participants) | 3 | 2 | 6
  Day 88 | 1.48 (0.623) | 1.01 (NA) — Insufficient samples were collected to assess SD. | 0.903 (1.17)
  Day 92: number analyzed (Participants) | 1 | 2 | 6
  Day 92 | 0.113 (NA) — Insufficient samples were collected to assess SD. | 0.00 (NA) — Insufficient samples were collected to assess SD. | 0.0953 (0.115)
  Day 99: number analyzed (Participants) | 4 | 2 | 6
  Day 99 | 0.00 (0.00) | 0.00 (NA) — Insufficient samples were collected to assess SD. | 0.110 (0.268)
  Day 113: number analyzed (Participants) | 3 | 2 | 5
  Day 113 | 0.00 (0.00) | 0.00 (NA) — Insufficient samples were collected to assess SD. | 0.00 (0.00)
  Day 127: number analyzed (Participants) | 4 | 2 | 6
  Day 127 | 0.00 (0.00) | 0.00 (NA) — Insufficient samples were collected to assess SD. | 0.00 (0.00)

7. Secondary Outcome: Phase 1b: Maximum Observed Serum Concentration (Cmax) of Efavaleukin Alfa
Time Frame: Day 1 (pre-dose) and 6 to 48 hours post-dose, and days 4, 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, Day 85 (pre-dose) and 6 to 72 hours post-dose, and days 92, 99, 113 and 127
Population: The PK analysis set: All participants who received at least one dose of Efavaleukin alfa and had at least one quantifiable PK sample collected. Only participants with PK data available for analysis are presented. Only cohorts with enrolled participants are included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 6 | 11 | 11
ng/mL
  First dose (Day 1) | 2.66 (0.852) | 23.0 (11.2) | 5.71 (5.10)
  Last dose (Day 85): number analyzed (Participants) | 4 | 2 | 6
  Last dose (Day 85) | 4.00 (2.05) | NA (NA) — Insufficient samples were collected to assess mean Cmax. | 3.22 (4.35)

8. Secondary Outcome: Phase 1b: Time to Maximum Observed Serum Concentration (Tmax) of Efavaleukin Alfa
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 6 | 11 | 11
hours
  First dose (Day 1) | 18 [12 to 24] | 24 [24 to 48] | 24 [12 to 72]
  Last dose (Day 85): number analyzed (Participants) | 4 | 2 | 6
  Last dose (Day 85) | 12 [12 to 12] | 30 [12 to 48] | 12 [6.0 to 24]

9. Secondary Outcome: Phase 1b: Area Under the Concentration-time Curve From Time 0 to 14 Days (AUC0-14) Post Dose
Description: AUC0-14 was only assessed for the participants who received Efavaleukin alfa using dosing schedule A.
Time Frame: Day 1 (pre-dose) and 6 to 48 hours post-dose, and days 4, 8, 11 and 15, Day 85 (pre-dose) and 6 to 72 hours post-dose, and days 92 and 99
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2
Number analyzed (Participants) | 6 | 10
hr*ng/mL
  First dose (Day 1) | 167 (60.9) | 1570 (859)
  Last dose (Day 85): number analyzed (Participants) | 4 | 2
  Last dose (Day 85) | 282 (207) | NA (NA) — Insufficient samples were collected to assess AUC0-14

10. Secondary Outcome: Phase 1b: Area Under the Concentration-time Curve From Time 0 to 7 Days (AUC0-7) Post Dose
Description: AUC0-7 was only assessed for the participants who received Efavaleukin alfa using dosing schedule B.
Time Frame: Day 1 (pre-dose) and 6 to 48 hours post-dose, and days 4 and 8, Day 85 (pre-dose) and 6 to 72 hours post-dose, and Day 92
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 10
hr*ng/mL
  First dose (Day 1) | 315 (239)
  Last dose (Day 85): number analyzed (Participants) | 6
  Last dose (Day 85) | 195 (264)

11. Secondary Outcome: Phase 1b: Number of Participants With Anti-Efavaleukin Alfa Binding Antibodies and Anti-Interleukin (IL-2) Binding Antibodies
Description: Number of participants who tested positive for anti-Efavaleukin alfa binding antibodies and number of those participants who cross-reacted with native human IL-2 (i.e. with anti-IL-2 binding antibodies) are reported.
Time Frame: Baseline up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: All participants who received at least 1 dose of investigational product and had a baseline and at least 1 post-baseline result. Only participants who tested positive for anti-Efavaleukin alfa antibodies were analyzed for presence of anti-IL2 binding antibodies. Only cohorts with enrolled participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 6 | 11 | 11
Participants
  Binding anti-AMG 592 antibody positive post-baseline with a negative or no result at baseline | 2 | 3 | 6 | 5
  Binding anti-IL2 antibody positive post-baseline with a negative or no result at baseline: number analyzed (Participants) | 3 | 3 | 8 | 5
  Binding anti-IL2 antibody positive post-baseline with a negative or no result at baseline | 0 | 0 | 1 | 1

12. Secondary Outcome: Phase 1b: Number of Participants With Anti-Efavaleukin Alfa Neutralizing Antibodies and Anti-IL-2 Neutralizing Antibodies
Description: The number of participants who tested positive for anti-Efavaleukin alfa neutralizing antibodies and number of participants with anti-IL2 neutralizing antibodies who tested negative or no result at baseline are reported.
Time Frame: Baseline up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: All participants who received at least 1 dose of investigational product and had a baseline and at least 1 post-baseline result. Only participants who tested positive for anti-Efavaleukin alfa antibodies were analyzed for presence of anti-IL2 neutralizing antibodies. Only cohorts with enrolled participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
Number analyzed (Participants) | 8 | 5 | 11 | 10
Participants
  Neutralizing anti-AMG 592 antibodies positive post-baseline with a negative or no result at baseline | 2 | 1 | 7 | 5
  Neutralizing anti-IL2 antibody positive post-baseline with a negative or no result at baseline: number analyzed (Participants) | 3 | 3 | 8 | 5
  Neutralizing anti-IL2 antibody positive post-baseline with a negative or no result at baseline | 0 | 0 | 1 | 1

13. Secondary Outcome: Phase 2a: Number of Participants Who Achieved an American College of Rheumatology 50 Percent Improvement Criteria (ACR 50) or 70 Percent Improvement Criteria (ACR 70) at Week 12
Description: ACR 50 and ACR 70 response defined as at least 50 percent or 70 percent improvement from baseline in both tender and swollen joint counts, and a 50 percent or 70 percent improvement or more in at least 3 of the following 5 criteria:
  * physician global assessment of disease activity (PGA)
  * subject global assessment of disease activity (SGA)
  * patient global assessment of joint pain
  * subject self-assessment of disability (HAQ-DI)
  * C-Reactive Protein (CRP)
Time Frame: Baseline and Week 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Phase 2a: Change From Baseline in Disease Activity Score (28 Joint) Calculated Using The Erythrocyte Sedimentation Rate Formula (DAS28-ESR) at Week 12
Description: Change from baseline in DAS28-ER at Week 12. DAS28-ESR was to assess disease activity in patients with rheumatoid arthritis. DAS28-ESR is a composite score that includes 4 variables: tender joint count (TJC) (based on 28 joints); swollen joint count (SJC) (based on 28 joints); participant's global assessment of health activity using 100 mm VAS: range 0 (no pain) to 100 (maximum pain imaginable); marker of inflammation assessed by ESR in mm/h. DAS28-ESR total score range from 0-10, higher score indicates more disease activity.
Time Frame: Baseline and Week 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Phase 2a: Change From Baseline in Disease Activity Score (28 Joint) Calculated Using the C-reactive Protein Formula (DAS-28-CRP) at Week 12
Description: Change from baseline in DAS28-CRP at Week 12. 2. DAS28-CRP was to assess disease activity in patients with rheumatoid arthritis. DAS28-CRP is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); participant's global assessment of health activity using 100 mm VAS: range 0 (no pain) to 100 (maximum pain imaginable); marker of inflammation assessed by CRP in mg/L. DAS28-CRP total score range from 0-10, higher score indicates more disease activity.
Time Frame: Baseline and Week 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase 2a: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were events with an onset after the administration of the first dose of study treatment.
  TEAEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Baseline up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Phase 2a: Number of Participants Who Experienced a Clinically Significant Change in Vital Signs
Description: as for outcome 2
Time Frame: Baseline up to Week 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Phase 2a: Number of Participants Who Experienced a Clinically Significant Change in Laboratory Safety Tests
Description: as for outcome 3
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Phase 2a: Efavaleukin Alfa Serum Concentration
Description: A summary of mean serum concentrations of Efavaleukin alfa over time.
Time Frame: Day 1 (pre-dose) and weeks 2, 4, 6, 8, 10 and 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Phase 2a: Maximum Observed Serum Concentration (Cmax) of Efavaleukin Alfa
Time Frame: Day 1 (pre-dose) and weeks 2, 4, 6, 8, 10 and 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Phase 2a: Time to Maximum Observed Serum Concentration (Tmax) of Efavaleukin Alfa
Time Frame: Day 1 (pre-dose) and weeks 2, 4, 6, 8, 10 and 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Phase 2a: Area Under the Concentration-time Curve (AUC) of Efavaleukin Alfa
Time Frame: Day 1 (pre-dose) and weeks 2, 4, 6, 8, 10 and 12
Population: No data is available for phase 2a. Study was terminated prior to any participants enrolling in phase 2a.
Arm/Group | Phase 2a: Placebo | Phase 2a: Efavaleukin Alfa
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-weeks double-blind treatment, 6-weeks safety follow-up)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Treatment emergent serious adverse events and other adverse events, including disease-related events are reported for all participants who received at least one dose of study drug.
  No data is available for phase 1b Cohort 4 or phase 2a cohorts as the study was terminated prior to any participants enrolling.
Arm/Group | Phase 1b: Placebo | Phase 1b: Efavaleukin Alfa Cohort 1 | Phase 1b: Efavaleukin Alfa Cohort 2 | Phase 1b: Efavaleukin Alfa Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/8 | 5/6 | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Placebo (N=8) | Phase 1b: Efavaleukin Alfa Cohort 1 (N=6) | Phase 1b: Efavaleukin Alfa Cohort 2 (N=11) | Phase 1b: Efavaleukin Alfa Cohort 3 (N=11)
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Placebo (N=8) | Phase 1b: Efavaleukin Alfa Cohort 1 (N=6) | Phase 1b: Efavaleukin Alfa Cohort 2 (N=11) | Phase 1b: Efavaleukin Alfa Cohort 3 (N=11)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Administration site reaction (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 4 | 2 | 3
Injection site hypersensitivity (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 6 | 8
Injection site swelling (General disorders) | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Administration related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Enrollment of the phase 1b part of this study was stopped as of 30 September 2019 due to data that suggested that there is not sufficient benefit-risk for the use of Efavaleukin alfa plus standard of care therapy in this study population. The study was terminated prior to the enrollment of any participants into phase 1b Cohort 4 and phase 2a cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03410056/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03410056/SAP_001.pdf